CLINICAL TRIAL: NCT05846698
Title: The Effects of Luo-Bu-Fu-Ke-Bi-RI Pill
Status: Completed | Type: Observational
Sponsor: Guoqing Zhou (Other)
Responsible Party: Sponsor-Investigator, Guoqing Zhou, associate chief physician, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: 2021-375
Record Dates: First submitted 2023-04-11; First posted 2023-05-06 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Climacteric Syndrome
MeSH Terms: interventions — tibolone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group
  Interventions: Drug: tibolone
- treatment group
  Interventions: Drug: Luo-Bu-Fu-Ke-Bi-RI Pill

INTERVENTIONS:
Drug: Luo-Bu-Fu-Ke-Bi-RI Pill — 10 pills twice daily
  Groups: treatment group
Drug: tibolone — 2.5 mg once daily
  Groups: control group

SUMMARY:
To investigate the effect of LBFKBRP on climacteric syndrome in women and explore its therapeutic mechanism.

ELIGIBILITY:
Clinical diagnosis of climacteric syndrome

Ages: 41 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: female
Sampling Method: Probability Sample
Enrollment: 276 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Sex hormone | 3 month

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No